CLINICAL TRIAL: NCT05742958
Title: The Quality of Recovery After Intrathecal Morphine or Adductor Canal Block Added to Spinal Anesthesia in Patients Undergoing Arthroscopic Anterior Cruciate Ligament Reconstruction
Brief Title: The Quality of Recovery After Intrathecal Morphine or Adductor Canal Block in Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Demet Laflı Tunay, Assist Prof, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cukurova Univ
Record Dates: First submitted 2023-02-05; First posted 2023-02-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Adductor Canal Block; Intrathecal Morphine; Arthroscopic Anterior Cruciate Ligament Reconstruction; Quality of Recovery
Keywords: intrathecal morphine; adductor canal block; quality of recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine (Group ITM) (Experimental): 12.5-15 mg hyperbaric 0.5% bupivacaine + 0.1 mg (0.1 mL) morphine with a single dose intrathecal injection through the L4-L5 interval (spinal anesthesia) + placebo adductor canal block (with 30 mL saline) will be administered.
  Interventions: Drug: Intrathecal morphine
- Adductor canal block (Group ACB) (Experimental): Spinal anesthesia from L4-L5 interval with 12.5-15 mg hyperbaric 0.5% bupivacaine + adductor canal block (30 mL 0.25% bupivacaine) will be applied.
  Interventions: Drug: Adductor canal block

INTERVENTIONS:
Drug: Intrathecal morphine — The study will be conducted in patients undergoing arthroscopic anterior cruciate ligament reconstruction surgery under spinal anesthesia. In this arm, 0.1 mg intrathecal morphine in addition to spinal anesthesia will be used for perioperative pain management. A placebo addctor canal block will also be performed for masking in these patients. The quality of recovery will be evaluated with a postoperative quality of recovery scale (QoR-40 questionnaire) at postoperative 24-hour and 14-day.
  Arms: Intrathecal morphine (Group ITM)
Drug: Adductor canal block — After providing complete sensory block in the lower extremities with spinal anesthesia, the thigh where the surgery will be performed will be brought into slight abduction and external rotation while the patient is in the supine position. The blockage of the saphenous nerve in the adductor canal will be performed with 30 mL of local anesthetic (0.25% bupivacaine) solution with a 22 gauge 5-8 cm long block needle from the mid-medial part of the thigh under ultrasound guidance. The quality of recovery will be evaluated with QoR-40 questionnaire at postoperative 24-hour and 14-day.
  Arms: Adductor canal block (Group ACB)

SUMMARY:
The Quality of Recovery 40 (QoR-40) is a multidimensional questionnaire that addresses many aspects of postoperative recovery. The QoR-40 has been used many times to measure the recovery of patients after different surgeries, and this questionnaire seems to be a reliable tool for evaluating anesthesia-related techniques, including regional anesthesia. Arthroscopic knee surgery causes moderate to severe postoperative pain for most patients. Various methods such as different systemic drugs, peripheral or central blocks and intra-articular injections have been developed for the effective, safe and long-term control of this pain. In recent years, it has been shown that regional anesthesia techniques reduce the need for opioids in orthopedic ambulatory surgeries and accelerate recovery and discharge. However, there is no consensus on which is the best approach among these various regional techniques. However, adductor canal block (ACB) and intrathecal morphine (ITM) are the preferred regional methods in the perioperative pain management of knee surgery. In this study, it was aimed to test the effectiveness of intrathecal morphine or adductor canal block added to spinal anesthesia on the quality of recovery in patients undergoing arthroscopic anterior cruciate ligament reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II adult patients aged 18-65 years undergoing elective arthroscopic anterior cruciate ligament reconstruction will be included in the study.

Exclusion Criteria:

* We will exclude patients with known coagulopathy, allergies to the studied drugs, obesity (BMI >35kg/m2), renal and/or hepatic insufficiency, chronic pain syndrome, mental impairment, depression, chronic alcoholism, and usage of antidepressant and analgesic drugs before surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
24-hour Quality of Recovery-40 (QoR-40) questionnaire scores | Postoperative 24-hour.
  The score ranges from 40 to 200. A higher score on the QoR-40 means better recovery following arthroscopic anterior cruciate ligament reconstruction.

SECONDARY OUTCOMES:
Numeric Rating Score (NRS) | Postoperative 1, 2, 4, 8, 12 and 24-hour.
  Numeric rating score for postoperative pain intensity. Pain intensity will be evaluated using a numeric rating scale with descriptive terms at intervals along a horizontal line of 10 cm length: 0 mm = no pain, 10 cm = worst pain imaginable.
Supplement analgesia requirement | Postoperative 1, 2, 4, 8, 12 and 24-hour.
  Amount of additional analgesics taken outside of the usual treatment protocol.
The time to first postoperative mobilisation | Duration of postoperative 24-hour
  Ambulation time
Discharge time | Duration of postoperative 24-hour
  Length of hospital stay
Treatment satisfaction | Postoperative 24-hour
  Treatment satisfaction will be assessed at 24 h using a 3-point rating scale ranging from 1 to 3: 1 = excellent satisfaction (Numeric Rating Score/NRS=0), 2 = good satisfaction (NRS=1-2), 3 = dissatisfaction (NRS=3-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant code, age, weight, height and information during surgery will be recorded. This information will not be shared with any person or organization.